CLINICAL TRIAL: NCT02546141
Title: Postprandial Plasma Amino Acid Concentrations After Dairy Consumption
Acronym: PARROT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL53912.081.15; METC nr 15/18 (Other: Medical Ethical Committee- Wageningen University)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Protein Digestion Kinetics
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- skimmed milk (UHT) (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: skimmed milk (UHT)
- skimmed milk (pasteurized) (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: skimmed milk (pasteurized)
- skimmed yoghurt (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: skimmed yoghurt
- full-fat milk (UHT) (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: full-fat milk (UHT)
- non-homogenized full-fat milk (pasteurized) (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: non-homogenized full-fat milk (pasteurized)
- full-fat cheese (semi-matured) (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: full-fat cheese (semi-matured)
- whey protein (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: whey protein
- micellar casein (Active Comparator): portion size that contains 25 g of protein, oral, single administration
  Interventions: Other: micellar casein

INTERVENTIONS:
Other: skimmed milk (UHT)
  Arms: skimmed milk (UHT)
Other: skimmed milk (pasteurized)
  Arms: skimmed milk (pasteurized)
Other: skimmed yoghurt
  Arms: skimmed yoghurt
Other: full-fat milk (UHT)
  Arms: full-fat milk (UHT)
Other: non-homogenized full-fat milk (pasteurized)
  Arms: non-homogenized full-fat milk (pasteurized)
Other: full-fat cheese (semi-matured)
  Arms: full-fat cheese (semi-matured)
Other: whey protein
  Arms: whey protein
Other: micellar casein
  Arms: micellar casein

SUMMARY:
This study was designed to obtain information about the change in postprandial amino acids in blood over time, after consumption of different dairy products, in an elderly population and how this relates to gastric emptying rate and feelings of satiety.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60y
* BMI 21-30 kg/m2
* Non-smoking
* Healthy as assessed by the NIZO lifestyle and health questionnaire
* Regular and normal Dutch eating habits as assessed by the NIZO lifestyle and health questionnaire (3 main meals per day)
* Veins suitable for cannulation (blood sampling)

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before Day 01 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome, including: Inflammatory bowel disease, hepatitis, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer
* Use of the following medication: glucose lowering drugs, insulin; medication that may impact gastric emptying (e.g. gastric acid inhibitors or laxatives)
* Diagnosed with diabetes, being treated for high blood glucose or increased fasting blood glucose (> 7 mmol/l in finger prick blood) as assessed during screening visit
* For men: Hb <8,5 mmol/l as assessed during screening visit; for women: Hb <7,5 mmol/l.
* Use of protein supplements
* Mental status that is incompatible with the proper conduct of the study
* A self-reported reported food allergy or sensitivity to dairy ingredients
* A self-reported allergy or sensitivity to acetaminophen
* Alcohol consumption > 28 units/week and 4/day
* Reported unexplained weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period
* Reported slimming or medically prescribed diet
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing or afraid to give up blood donation during the study
* Personnel of NIZO food research or Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results and eventual adverse events to and from his general practitioner

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
iAUC for postprandial individual plasma amino acids | 0-300 min after consumption
Cmax for postprandial individual plasma amino acids | 0-300 min after consumption
Tmax for postprandial individual plasma amino acids | 0-300 min after consumption

CONTACTS AND LOCATIONS:
Locations (1):
- NIZO food research, Ede, Netherlands